CLINICAL TRIAL: NCT03515252
Title: A Phase I Study to Evaluate the Safety and Efficacy of Autologous Immune Killer Cells in Patients With Late Stage Hepatocellular Carcinoma or Lung Cancer
Brief Title: Study of Autologous Immune Killer Cells in Patients With Late Stage Hepatocellular Carcinoma or Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ivy Life Sciences, Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVY 01
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IV; Hepatocellular Carcinoma by BCLC Stage; Lung Cancer; Liver Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Late stage lung cancer and liver cancer (Experimental): Immune Killer Cells (IKC)
  Interventions: Biological: Immune Killer Cells (IKC)

INTERVENTIONS:
Biological: Immune Killer Cells (IKC)

SUMMARY:
This is a phase I clinical study. Blood is drawn from the patient and brought to our laboratory for isolation of immune cells. These immune cells are then proliferated over a two week period and used to produce our patented product IKC (Immune Killer Cells). The IKC will then infused back into the patient to treat the cancer. Each patient will receive a total of six infusions.

DETAILED DESCRIPTION:
This is a phase I clinical study. Blood is drawn from the patient and brought to our laboratory for isolation of immune cells. These immune cells are then proliferated over a two week period and used to produce the patented product IKC (Immune Killer Cells). The IKC will then infused back into the patient to treat the cancer. Each patient will receive a total of six infusions.

For each indication (cancer of the lung or liver) 10 patients are anticipated to be recruited, making a total of 20 subjects. All subjects will receive treatment as this is a single-arm study.

ELIGIBILITY:
Inclusion Criteria:

1. subjects had voluntarily given written informed consent
2. subjects had CT scan on lung or liver tumors within the past 4 weeks of the screening visit
3. subjects who were histologically or pathologically confirmed with locally advanced or metastatic lung cancer or HCC
4. subjects who did not have valid therapy, ever failed with other therapy, or refused or were not appropriate for other therapies for lung cancer or HCC
5. subjects' ECOG performance status ≤ 2
6. subjects with life expectancy ≥ 3 months

Exclusion Criteria:

1. subjects with medical history of gout
2. subjects who had participated other clinical trials within 4 weeks before the screening visit
3. subjects with positive result of HIV or HTLV test within 4 weeks before the screening visit
4. subjects with clinically significant diseases other than cancer
5. subjects with myocardial infraction, stroke, or congestive heart failure within 3 months before the screening visit
6. female subjects who were pregnant or lactating or women of child-bearing potential but unable to take adequate contraception
7. subjects with history of alcohol, drug or other substance abuse
8. subjects with disease of bacteremia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04-26 (Actual); Primary Completion 2006-11-02 (Actual); Study Completion 2007-06-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 5 months
  Adverse Events (AE) and Serious Adverse Events (SAE) will be recorded and evaluated for their relationship to the treatment

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) | 4 months
  Record net changes of tumor sizes
Quality of Life (QOL) | 5 months
  The assessment will be performed using The World Heath Organization Quality of Life Questionnaire (WHOQOL)
  This questionnaire produces a quality of life profile. It is possible to derive four domain scores. The four domain scores denote an individual's perception of quality of life in each particular domain (1. Physical health 2. Psychological 3. Social relationships 4. Environmental) Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
  The mean score of items within each domain is used to calculate the domain score (min: 0 max: 100)
  Domain scores are then calculated (divide domain score by 4) to produce a final QOL Score (i.e. higher scores denote higher quality of life min: 0 max:100).

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Ching Yang, MD, PhD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital